CLINICAL TRIAL: NCT02527642
Title: Commercial Single Step (Vitrolife -G-TL™) Media Compared With Cornell Media: A Randomized Controlled Trial by Time-Lapse System- Single Step vs Sequential Media
Brief Title: Commercial Single Step (Vitrolife -G-TL™) Media Compared With Cornell Media
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Vitrolife (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1411015635
Record Dates: First submitted 2015-07-28; First posted 2015-08-19 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CRM sequential media (C1/C2) (Active Comparator): CRM sequential media, formulated according to the stages of embryo development, is used to culture the embryos from oocyte fertilization to blastocyst stage.
  Interventions: Other: embryo culture in buffered media
- CRM single step media (C3) (Active Comparator): CRM single step media is used to culture the embryos from oocyte fertilization to blastocyst stage.
  Interventions: Other: embryo culture in buffered media
- Vitrolife media G1/2 Sequential (Experimental): Vitrolife sequential media, formulated according to the stages of embryo development, is used to culture the embryos from oocyte fertilization to blastocyst stage.
  Interventions: Other: embryo culture in buffered media
- Vitrolife G-TL Time Lapse media Single Step (Experimental): G-TL Time Lapse Single step (time lapse) media is formulated for continuous culture from oocyte fertilization to blastocyst stage.
  Interventions: Other: embryo culture in buffered media

INTERVENTIONS:
Other: embryo culture in buffered media — compare media that supports human embryo development in the laboratory (in vitro) using Time-Lapse system.
  Other Names: Embryo media- CRM media vs Vitrolife

SUMMARY:
This is a randomized, controlled, single-center study in otherwise healthy infertile female subjects undergoing in vitro fertilization (IVF). The subjects recruited for this study will be among those patients who have been diagnosed with infertility and are planning to undergo IVF at the centers where this study is being performed. The patients will have undergone the usual informed consent procedure at the center.

DETAILED DESCRIPTION:
Subjects will undergo ovarian stimulation, oocyte retrieval, IVF, and Intra Cytoplasmic Sperm Injection (ICSI) procedure following the center's usual procedures. The cohort of injected oocytes from each patient will be randomly divided between the one step and sequential medias: CRM (Cornell- Center for Reproductive Medicine) media (C1/C2 or C3) vs G-TL Time Lapse media or G-1/G-2 media. Single step or sequential media are both buffered mediums for culture from oocyte fertilization to blastocyst stage. Sequential media is formulated according to the stages of embryo development and embryos are re-cultured in medias according to their stage of development. Single step (time lapse) media is formulated for continuous culture from D0 to Day 5/6.

Mature oocytes will be randomized via a non-bias computer program into two to four of the study groups: G-TL commercial single step (Vitrolife), Vitrolife's sequential media, Cornell's single step , and Cornell's sequential media. Oocytes will be divided randomly among the various media dependent upon the number of mature oocytes. I.e.: 10 oocytes injected = 2 media groups; 15 oocytes injected = up to 3 media groups; 20 oocytes injected = up to 4 media groups.

"Best grade" embryos will be transferred regardless of media source. If embryos are transferred from multi-source media and if researchers are unable to determine the media source after transfer, the subject will not be included in the outcome data portion of the study- e.g pregnancy outcome.

The Time-Lapse monitoring system will be used as standard clinical practice to observe development and document timing of embryo cleavages and morphology dynamics.

Endpoints will be Day 3 and Day 5/6 embryo development, implantation and pregnancy rate. The study is approximately 2 months, the estimated time it takes a physician to perform one IVF-ART IVF- Assisted Reproductive Technology) treatment cycle. If embryos are frozen, the patient may be in the study until the time they choose to thaw the embryos or up to 1 year if they become pregnant.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age or younger (maternal) 65 years of age or younger (paternal)
* Patient must have 10 or greater than 10 mature oocytes, ICSI only
* Fresh or frozen (including donor) sperm can be used. Fresh oocytes only (including donor)
* Frozen embryos from this study can be included in the outcome portion of this study.
* Single or double Blastocyst transfer only

Exclusion Criteria:

* Patients having PGS (Pre-implantation Genetic Screening)
* 3 or more previous failed cycles
* Sperm obtained by testicular biopsy
* Previous enrollment in the study
* Non blastocyst transfer
* Co-culture patients
* Outcome data portion exclusion only:

Multi-source media transfers if researchers are unable to determine the media source after transfer.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2015-07; Primary Completion 2016-10-17 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Embryo development | 1 year
  Comparison of embryo development using standard assessments of morphokenetics of embryo development

SECONDARY OUTCOMES:
Embryo transfer rate | 1 year
  Percentage of embryo transferred in each arm.
Clinical pregnancy rates | within 3 months of embryo transfer
  Percentage of embryos transferred that implant into the uterus by evidence of a fetal sac by ultrasound

OTHER OUTCOMES:
Number of participants pregnant after Frozen Embryo Transfer | 2 years
  Pregnancy rate from frozen embryo transfer in each arm.

CONTACTS AND LOCATIONS:
Overall Officials: Nikica Zaninovic, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Center fo Reproductive Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No